CLINICAL TRIAL: NCT04706520
Title: A Randomized, Double-Blinded, Placebo-Controlled Study to Assess the Effects of Chronic Consumption of Vinegar on Visceral Adiposity in Overweight Adults
Brief Title: Chronic Consumption of Vinegar on Visceral Adiposity in Overweight Adults (VAnish)
Acronym: VAnish
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: study sponsor ended due to recruitment issues
Sponsor: Pennington Biomedical Research Center (Other)
Collaborators: Mizkan Holdings Co., Ltd. (Industry)
Responsible Party: Principal Investigator, John Apolzan, Assistant Professor, Director Clinical Nutrition and Metabolism Lab, Pennington Biomedical Research Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PBRC-2020-048
Record Dates: First submitted 2021-01-07; First posted 2021-01-13 (Actual); Last update posted 2021-11-16 (Actual); Status verified 2021-11

CONDITIONS: Body Composition

STUDY DESIGN:
Intervention Model Description: VAnish is a randomized, placebo-controlled, parallel study model with 3 groups consisting of 20 participants who will all consume 2 bottles of study product per day. Group 1 will receive 400mL/day of vinegar; Group 2 will receive 200mL/day of vinegar and 200mL/day of the placebo drink; Group 3 will receive 400mL/day of the placebo drink.
Who Masked: Participant, Investigator
Masking Description: Participants will be blinded as to which group they are randomized since both the vinegar and placebo beverages are the same in appearance and taste. The Investigators, clinic staff, and intervention staff are also all blinded. The only unblinded group is the Metabolic Kitchen who facilitates randomization and distribution of study product.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1: Vinegar (Experimental): Participants will consume 400 mL/day vinegar beverage providing 1,500 mg/day acetic acid [200 mL vinegar beverage, twice per day (prior to breakfast and dinner)] for 12 weeks.
  Interventions: Dietary Supplement: Study Beverage Consumption
- Group 2: Vinegar/Placebo Combination (Experimental): Participants will consume 200 mL/day vinegar beverage and 200 mL/day placebo beverage providing 1,200 mg/day lactate [200 mL placebo beverage 1x/day] and 750 mg/day acetic acid [200 mL vinegar beverage 1x/day] (prior to breakfast and dinner) for 12 weeks.
  Interventions: Dietary Supplement: Study Beverage Consumption
- Group 3: Placebo (Placebo Comparator): Participants will consume 400 mL/day placebo beverage containing 1,250 mg/day lactate [200 mL placebo beverage, and 200 mL placebo beverage (prior to breakfast and dinner) for 12 weeks.
  Interventions: Dietary Supplement: Study Beverage Consumption

INTERVENTIONS:
Dietary Supplement: Study Beverage Consumption — All participants will follow the same intervention as the study staff is blinded in addition to the participant. Randomized participants will be asked to consume 2 bottles per day of a study beverage for 12 weeks. Compliance checks will occur remotely by having participants send photos of their bottles each day and weekly phone/video calls with intervention staff. Participants will be asked to keep their diet and activity level consistent throughout the 12 weeks.

SUMMARY:
To assess, relative to a placebo, the effects of consuming 400 mL/day or 200 mL/day of a vinegar beverage providing either 1,500 mg/day of acetic acid (in two 200 mL doses daily) or 750 mg/day of acetic acid (in one 200 mL dose daily), respectively, for 12 weeks on VAT (MRI). Thus the 2 active comparator arms 400 mL and 200 mL of vinegar will be independently tested compared to placebo.

DETAILED DESCRIPTION:
It has been reported that increased visceral adipose tissue (VAT) is associated with a range of metabolic abnormalities, including decreased glucose tolerance and insulin sensitivity, as well as adverse lipid profiles, all of which are risk factors for type 2 diabetes and CVD (WHO, 2008). In the European Union, a sustained reduction in abdominal fat, and in particular visceral fat, is considered a beneficial physiological effect for adults with adverse health effects associated with excess abdominal fat, including impaired glucose tolerance, dyslipidemia, and hypertension (EFSA, 2012).

This clinical trial is a randomized, double-blinded, placebo-controlled, parallel, single-center study involving a total of 60 male and female adults (aged 18 to 60 years, inclusive) who are overweight (BMI between 25.0 to ˂30.0 kg/m2) and have abdominal obesity (waist circumference >102 cm for males, >88 cm for females) (ATP III, 2001). Each subject's duration of participation will be a total of ~14 weeks, including a ~2-week screening visit and a ~12-week randomized placebo-controlled double-blinded supplementation period.

On the first day of the ~2-week screening period (~Day -14), subjects will be screened according to the study inclusion and exclusion criteria. Subjects meeting all of the inclusion criteria and none of the exclusion criteria will be invited to return to the clinic for a second screening visit (~Day -7). During this second screening visit, subjects will be instructed on how to use the Fitbit (accelerometer) and on how to properly complete the food intake diary. Subjects will be instructed not to alter their dietary intakes or their physical activity levels during the subsequent week, and to record the information as accurately as possible. Participants will be asked to record at least 3 days of physical activity and dietary measurements that includes at least 1 weekend day. Subjects will then be instructed to return to the clinic ~1 week later for the collection of baseline measures (Day 0).

Following the collection of baseline measures on Day 0, subjects will be randomized to the placebo or one of the vinegar groups. Each group will consist of 20 subjects. Randomization will be adaptive according to sex and age; subjects will be asked to return to the clinic twice, once ~11 weeks after the baseline visit to obtain food intake diary, accelerometer, and stool collection materials, and again, ~12 weeks after the baseline visit (i.e., 12 weeks after the baseline visit). Each subject will be required to make a total of 4 visits to the clinical research site (i.e., Days -14, -7, 0, and 84). The entire duration of the clinical study is expected to be approximately 52 weeks from subject enrollment to study closeout.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females between 18 and 60 years of age (inclusive) of any ethnicity, free of medications except for oral contraceptives (see inclusion criterion 8).
2. Subjects are overweight at screening (Visit 1, Day -14), as defined by a BMI of between 25.0 to ˂30.0 kg/m2, inclusive.
3. Subjects have abdominal obesity at screening (Visit 1, Day -14), as defined by a waist circumference of >102 cm for males or >88 cm for females (ATP III, 2001).
4. Physical examination and vital signs are normal, or deemed abnormal but clinically insignificant by the Principle and/or Medical Investigator.
5. Clinical laboratory evaluations (including but not limited to clinical chemistry [fasted at least 8 hours], including creatine phosphokinase (CPK)], amylase, lipid profile, thyroid stimulating hormone (TSH), free thyroxine (T4), cortisol) complete blood count (CBC), are within the reference ranges for the central laboratory, unless deemed not clinically significant by the Investigator.
6. Males who are sterile or agree to use an approved method of contraception, with an approved method of contraception considered a barrier method (diaphragm, cervical cap, or condom) plus a contraceptive jelly (spermicidal foam, gel, film, cream, or suppository). If the female sexual partner of the male is using an approved form of contraception (see inclusion criterion 8), the male is not required to be sterile or, if not sterile, to use an approved form of contraception.
7. Female subjects who are postmenopausal (absence of menses for 1 year or more), women who are surgically sterilized, or women of child-bearing potential (WOCBP) who are nonlactating and have been using an effective form of birth control for a minimum of 6 months prior to screening and agree to continue using the effective form of birth control during the study and for 30 days after the treatment period [effective forms of birth control include oral pills with a concentration of at least 50 μg of the estrogenic component of a biphasic or triphasic pill; transdermal, injectable, or implantable contraceptive; intrauterine device; or double-barrier method (e.g., diaphragm and condom). Abstinence is not considered an acceptable form of birth control.] WOCBP who are using low dose oral birth control must also use a barrier method of contraception for the duration of the study.
8. Subjects who, during the investigative period, are willing to:

   1. Consume the prescribed amount of vinegar beverage;
   2. Wear the accelerometer (Fitbit);
   3. Complete food intake diary as required.
   4. Collect stool sample
   5. Willing to archive blood and stool samples
9. Subjects who are capable of giving informed consent and complying with all study procedures/ requirements.

Exclusion Criteria:

1. Subjects who, in the past 6 months, have dieted or have used any supplement/medication intended to affect body weight or suppress appetite
2. Subjects with a history of an eating disorder in the last 5 years.
3. Subjects who have had or are planning to have bypass surgery, stomach banding surgery, or any other surgical procedure(s), including those of a cosmetic nature, that attempt to aid/promote weight loss or alter body composition.
4. Subjects with Type I or Type 2 diabetes mellitus.
5. Subjects with endocrine disease (thyroid dysfunction defined by serum levels of T4, TSH or a past diagnosis of Cushing syndrome).
6. Subjects who have a history or presence of significant pulmonary, hepatic, renal, hematological, gastrointestinal, endocrine, immunological (e.g., HIV/AIDS), dermatologic, urological, neurological, psychiatric, or cardiovascular disease or disorder.
7. Subjects with any implanted electric device (such as a cardiac defibrillator) or other medical device that would allow for them to perform an MRI.
8. Women with polycystic ovarian syndrome.
9. Women who began taking oral contraceptives or hormone replacement therapy recently, within the last 6 months.
10. Women who plan to become pregnant during the study or were pregnant or nursing within the past year.
11. Subjects who have recently undergone barium tests/exams (within 7 days), or who have had a nuclear medicine scan or injection with an x-ray dye (within 3 days).
12. Subjects who have a history or presence of alcoholism or drug abuse within the previous 2 years and/or a positive urine drug screen at screening.
13. Subjects who have quit smoking in the last 6 months or who plan on quitting/altering smoking habits during their participation in this clinical trial.
14. Subjects who donated 1 pint or more of blood or blood products within 56 days prior to the study, and/or had a plasma donation within 7 days prior to the study or who plan to donate blood or blood products during their participation in this clinical trial.
15. Subjects with poor peripheral venous access that would preclude blood collection.
16. Subjects who are currently participating or plan to participate in any other investigational trial in which receipt of an investigational product will occur.
17. Subject who resides in the same household as another subject already participating in the study.
18. Subjects who have any condition that would make them, in the opinion of the Investigator, unsuitable for the study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2021-02-10 (Actual); Primary Completion 2021-11-04 (Actual); Study Completion 2021-11-04 (Actual)

PRIMARY OUTCOMES:
Visceral Adipose Tissue (VAT) | 12 weeks
  The primary objective is to assess the effects of consuming vinegar (1500mg/day and 750mg/day) on visceral adipose tissue via MRI as compared to a placebo.

SECONDARY OUTCOMES:
Body Weight | 12 weeks
  A secondary outcome is to assess, relative to a placebo, the effects of consuming vinegar (1500mg/day and 750 mg/day) on body weight.
Triglycerides | 12 weeks
  A secondary outcome is to assess, relative to a placebo, the effects of consuming vinegar (1500mg/day and 750 mg/day) on triglycerides.

CONTACTS AND LOCATIONS:
Overall Officials: Frank J Greenway, MD, Principal Investigator — Pennington Biomedical Research Center; Shengping Yang, PhD, Principal Investigator — Pennington Biomedical Research Center
Locations (1):
- Pennington Biomedical Research Center, Baton Rouge, Louisiana, United States

IPD SHARING:
Plan to Share IPD: No